CLINICAL TRIAL: NCT07085130
Title: Comparison of the Effects of Cold Application and Exercise With Virtual Reality Interventions on Pain, Kinesiophobia, and Fragility Levels in Patients With Diabetic Peripheral Neuropathy
Brief Title: The Effect of Hand and Foot Exercises Combined With Cold Application or Virtual Reality on Diabetic Neuropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva SERT, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAU-hand and foot exercises
Record Dates: First submitted 2025-07-11; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetic peripheral neuropathy; hand and foot exercises; cold application; virtual reality; kinesiophobia; fraility; neuropatic pain
MeSH Terms: conditions — Kinesiophobia | interventions — Exercise; Exergaming

STUDY DESIGN:
Intervention Model Description: In terms of the reliability of the study results, patients in this study will be divided into groups using a stratified randomization method. Patients will be randomly assigned to two intervention (I) and one control (C) groups according to their age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention: Cold Application (Experimental): Patients in the cold application intervention group will be evaluated during the first week and data collection forms will be completed. They will perform the hand and foot exercises in the exercise video three days a week, after which cold compress bags will be applied to their hands and feet for 5-10 minutes. They will be cooled to -25 to -30 °C for at least 3 hours before use.
  Interventions: Behavioral: Exercises and cold application
- Intervention: Virtual Reality (Experimental): Patients in the virtual reality intervention group will be evaluated during the first week and data collection forms will be completed. The virtual reality application will be taught through explanation and demonstration. The researcher will accompany the patients and the glasses and headphones will be put on the patient in a comfortable sitting position. As part of the application, patients will attempt to perform hand and foot exercises for an average of 15 minutes in a virtual environment accompanied by snowy landscapes and snow-themed sounds. The patient will be observed by the researcher during the application, and if symptoms such as dizziness, headache, or discomfort occur during the virtual reality application, the application will be terminated. Patients in the virtual reality intervention group will perform the virtual reality application three times a week for eight weeks. Patients will record their virtual reality applications in the Virtual Reality Application Diary.
  Interventions: Other: Exercises and virtual reality
- Control (No Intervention): Patients in the control group will be allocated time similar to the intervention flow applied to the intervention groups, and diabetic peripheral neuropathy will be explained. In this context, the control group patients will be evaluated in the first week, data collection forms will be filled out, and neuropathy management training will be explained by the researcher. The content of the presentation will cover the treatment and management of diabetic neuropathy.
- Intervention: Hand and foot exercises (Experimental): In this study, hand and foot exercises will be combined with both cold application and virtual reality, and both intervention groups will perform these exercises. Patients will perform hand and foot exercises approximately three times a week for about 15 minutes. Hand and foot exercises are an easy-to-perform, low-cost type of exercise designed to relieve individuals who experience numbness and tingling-like pain. Patients will perform hand movements such as the snail movement, making a full and half fist, the claw movement, and rolling a ball. For foot exercises, they will perform movements such as crumpling a towel, rolling a ball, and spreading the toes.
  Interventions: Behavioral: Exercises and cold application; Other: Exercises and virtual reality

INTERVENTIONS:
Behavioral: Exercises and cold application — Hand and foot exercises combined with cold application interventions are non-pharmacological methods used to reduce pain, kinesiophobia, and fragility levels in patients with diabetic peripheral neuropathy.
  Other Names: cold application; hand and foot exercises
  Arms: Intervention: Cold Application; Intervention: Hand and foot exercises
Other: Exercises and virtual reality — Performing hand and foot exercises in a cold, snowy virtual environment using virtual reality goggles may be a non-pharmacological intervention to alleviate burning-type hand and foot pain in patients with diabetic neuropathy.
  Other Names: virtual reality; hand and foot exercises
  Arms: Intervention: Hand and foot exercises; Intervention: Virtual Reality

SUMMARY:
The study will be conducted to determine the effect of cold application and virtual reality (VR) or combined hand and foot exercises on pain intensity, kinesiophobia, and fragility levels in patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetic neuropathy is associated with high morbidity and mortality rates in both Type 1 and Type 2 diabetes patients, increasing the risk of foot ulcers and amputations, hospital admission rates, and healthcare costs. It also causes a decline in individuals' quality of life, functional capacity, and physical activity levels. Especially at night, increased pain disrupts individuals' sleep patterns; psychological problems such as stress, anxiety, and depression are common. Diabetic neuropathy is a complication that affects individuals physically, psychologically, and socially. It is known that neuropathic pain accompanies the clinical picture in 25-50% of patients with diabetic neuropathy. One of the exercise programs used by healthcare professionals to alleviate symptoms in patients with peripheral neuropathy is hand and foot exercises. Studies in the literature show that hand and foot exercises performed by patients with peripheral neuropathy reduce pain levels, improve quality of life, and increase physical activity levels.Another alternative method used in the treatment of neuropathic pain is cold application. Cold application causes vasoconstriction in the blood vessels in the area where it is applied, slowing down tissue metabolism. In diabetic peripheral neuropathy, patients often describe a burning sensation in their hands and feet. Virtual reality technology has been used in the treatment and care of many diseases in the healthcare sector in recent years. VR is known to be quite effective in reducing pain, managing symptoms, and continuing care and rehabilitation outside of the hospital. VR applied to patients with diabetic peripheral neuropathy generally involves exercise interventions.

The study population will consist of patients with diabetic peripheral neuropathy who visit the Diabetes Clinic of the Department of Internal Medicine at Sakarya University Education and Research Hospital. All patients who meet the inclusion criteria will be included in the study population. The G*Power 3.1.9.2 program was used to calculate the number of individuals to be sampled. In this regard, a power level of 90% and a significance level of 0.05 were accepted in calculating the research sample. The power analysis is based on a previously published article that addressed a similar topic and provided mean and standard deviation values (Elshinnawy et al., 2024). According to the calculations, 42 patients (14 individuals in each group) are planned to be included in the study sample.The study will use a socio-demographic form, a neuropathic pain assessment questionnaire (DN4), the Tampa Kinesiophobia Scale, and the Tilburg Frailty Scale.

The study will consist of two intervention groups and one control group. The Cold Application group will perform the hand and foot exercises in the exercise video three days a week, then apply cold compress bags to their hands and feet for 5-10 minutes. Patients in the virtual reality group will exercise for 15 minutes with a hand and foot exercise video in a virtual environment accompanied by cold-themed sounds and the sound of snow.Patients in the control group will be allocated time similar to the intervention flow applied to the intervention groups, and diabetic peripheral neuropathy will be explained. The explanation will cover the treatment and management of diabetic neuropathy. Patients will perform this exercise for eight weeks, and at the end of eight weeks, individuals' pain, kinesiophobia, and fragility will be assessed.

No studies have been found in the literature where hand and foot exercises were applied to patients with diabetic neuropathy in combination with VR or cold application. In our study, hand and foot exercises are planned to be applied to patients in both the cold application and virtual reality intervention groups. This will ensure that patients feel relaxed after exercise and that multiple non-pharmacological methods are used simultaneously. As a result of all these interventions, patients' pain levels and kinesiophobia will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Those who volunteer to participate in the study

* Those who have been diagnosed with diabetes at least 6 months ago
* Those who show symptoms of neuropathy
* Those over the age of 18
* Those without cognitive or psychiatric diagnoses
* Those who are open to communication and cooperation
* Those who use a smartphone

Exclusion Criteria:

* Those with neurological disorders other than neuropathy
* Those with any additional orthopedic or systemic disorders that would prevent them from performing the exercises
* Those who have had a lower extremity pathology (surgery, fracture, soft tissue injury, etc.) in the past 6 months
* Those who are pregnant during the study period
* Those who wish to withdraw from the study of their own accord

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Changes in kinesiophobia | At the end of eight weeks
  As a result of the intervention, the Tampa Kinesiophobia Scale will be used to evaluate the differences and effects between the intervention and control groups in terms of fear of movement levels. The Turkish validity and reliability study of the scale developed by Miller and colleagues (1991) was conducted by Yılmaz and colleagues (2011). The TKÖ is a 17-item scale developed to measure fear of movement/re-injury. Each question in the scale uses a 4-point Likert scale (1 = Strongly disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Strongly agree). The total score obtained from the questionnaire ranges from 17 to 68. A high score on the scale indicates a high level of kinesiophobia.
Change in the neuropathic pain levels | at the end of eight weeks
  Following an eight-week intervention, the Douleur Neuropathique en 4-DN4 questionnaire will be used to assess whether there has been a reduction in patients' neuropathic pain levels. The DN4 pain questionnaire, developed by a neuropathic pain group, consists of four questions that inquire about the characteristics, type, location, and aggravating factors of neuropathic pain. According to the scale, neuropathic pain is assessed with a total of four questions, the first two of which are based on direct interviews with the patient and the last two on the patient's clinical examination. The Turkish validity and reliability study was conducted by Ünal Çevik and colleagues (2010). The questions in the questionnaire are answered with "yes" or "no." Each 'yes' answer is scored as 1 point, and each "no" answer is scored as 0 points. According to the scale, the threshold value for neuropathic pain is set at 4/10 or higher.
Change in fraility | At the end of eight weeks
  As a result of the intervention, the fragility levels of patients with diabetic peripheral neuropathy will be assessed using the Tilburg Fraility Scale. The Turkish validity and reliability study of the scale developed by Gobbens and colleagues (2010) was conducted by Arslan and colleagues (2018). The TKÖ consists of 15 questions and 3 sub-dimensions that assess vulnerability. The scale includes 8 questions that assess the physical domain, 4 questions that assess the psychological domain, and 3 questions that assess the social domain. Eleven items of the TKÖ are evaluated in two categories: "Yes" and "No." Four items of the TKÖ are scored as "yes," "sometimes," and "no." The total score that can be obtained from the scale ranges from 0 to 15, with scores of 5 and above indicating the presence of vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: Busra Gurcay, Research Assistant, Principal Investigator — Sakarya University Health Science Institute
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No